CLINICAL TRIAL: NCT06769113
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX43 (Anti-PD-L1 ADC) in Patients With Recurrent/Metastatic Esophageal Squamous Cell Carcinoma (ESCC) Failed or Intolerance to Standard First-line Therapy
Brief Title: A Phase II Clinical Study to Evaluate HLX43 in Patients With Recurrent/Metastatic ESCC Failed or Intolerance to Standard Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX43-ESCC201
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HLX43 DOSE 1 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 DOSE 1
- HLX43 DOSE 2 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 DOSE 2
- HLX43 DOSE 3 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 DOSE 3

INTERVENTIONS:
Drug: HLX43 DOSE 1 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 DOSE 1
Drug: HLX43 DOSE 2 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 DOSE 2
Drug: HLX43 DOSE 3 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 DOSE 3

SUMMARY:
The study is being conducted to explore the reasonable dosage and evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in Patients with Recurrent/Metastatic Esophageal Squamous Cell Carcinomar (ESCC) Failed or Intolerance to Standard First-Line Therapy.

DETAILED DESCRIPTION:
This study is an open-label phase II clinical study to explore the reasonable dosage and evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in Patients with Recurrent/Metastatic Esophageal Squamous Cell Carcinomar (ESCC) Failed or Intolerance to Standard First-Line Therapy.

In this study, eligible subjects will be randomized at 1:1:1 ratio, and the patients will be administered with HLX43 at different doses via intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research; To fully understand and understand this study and to sign the Informed Consent Form (ICF); Willing to follow and able to complete all test procedures;
2. The age of signing ICF is ≥ 18 years old and ≤ 75 years old;
3. Esophageal Squamous Cell Carcinoma (ESCC) confirmed by histopathology or cytology;
4. Patients with advanced esophageal squamous cell carcinoma who have failed or are intolerant to prior first-line standard therapy (for patients with PD-L1 expression positive [CPS ≥1], first-line standard therapy is defined as platinum-based chemotherapy and immune checkpoint inhibitor [ICI] therapy; for patients with PD-L1 expression negative [CPS <1], first-line standard therapy is defined as platinum-based chemotherapy). Intolerable toxicity refers to the occurrence of CTCAE grade ≥3 adverse events.;
5. Within 4 weeks prior to the first administration of the medication, at least one measurable target lesion must be evaluated according to the RECIST v1.1 criteria;
6. Tumor tissue should be provided as much as possible for an evaluable PD-L1 expression result at Screening period；
7. Before the initial administration of the study drug, there should be at least a 3-week interval or 5 times the half-life of the last cytotoxic chemotherapy, immunotherapy, or biological therapy, whichever is shorter. There should be at least a 2-week interval from the previous small molecule targeted therapy, at least a 1-week interval from traditional Chinese medicine treatment with antitumor indications or minor surgery. Additionally, treatment-related adverse events (AEs) should have recovered to NCI-CTCAE grade ≤ 1 (except for grade 2 peripheral neurotoxicity and alopecia)；
8. The ECOG physical performance score of 0-1 in the week prior to randomization；
9. Expected survival ≥ 3 monthes；
10. Laboratory tests within the previous week confirm adequate organ function (within 14 days prior to the first dose of medication, without receiving interventions such as blood transfusions, granulocyte colony-stimulating factor, or recombinant human thrombopoietin)；
11. Male and female subjects of childbearing potential must agree to use at least one highly effective method of contraception during the trial and for at least 6 months after the last dose of the study drug. Female subjects of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.

Exclusion Criteria:

1. History of any second malignant tumor within the first 2 years prior to randomization;
2. BMI <17.5 kg/m2；
3. Symptomatic, untreated, or progressively worsening central nervous system (CNS) or leptomeninges metastases;
4. After appropriate intervention, uncontrollable pleural effusion, pericardial effusion or ascites still need to be drained frequently;
5. A history of ≥ grade 3 radiation pneumonia; A history of (non-infectious) interstitial lung disease (ILD) requiring steroid use, or a current ILD, or suspected ILD cannot be ruled out by imaging at the time of screening; Or there are lung diseases leading to clinical severe respiratory impairment;
6. Subjects exhibit poorly controlled cardiovascular clinical symptoms or diseases, including but not limited to: (1) NYHA class II or above heart failure, or left ventricular ejection fraction (LVEF) < 50%; (2) unstable angina; (3) myocardial infarction or cerebrovascular accident within the last 6 months (excluding lacunar infarction, minor ischemic stroke, or transient ischemic attack); (4) uncontrolled arrhythmias (including QTc interval ≥ 450 ms for males, ≥ 470 ms for females) (QTc interval calculated by Fridericia's formula); (5) poorly controlled hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg despite active treatment);
7. Subjects who are preparing for or have previously received an organ or bone marrow transplant;
8. Within the 2 weeks prior to randomization, there is the presence of an active systemic infectious disease requiring intravenous antibiotic treatment;
9. Used strong inhibitors or strong inducers of CYP2D6 or CYP3A within 2 weeks prior to randomization;
10. Received systemic corticosteroids (prednisone >10 mg/day or an equivalent dose of similar drugs) or other immunosuppressive treatments within 14 days prior to the first dose; with the following exceptions: use of topical, ophthalmic, intra-articular, intranasal, and inhaled corticosteroids; short-term use of corticosteroids for prophylactic treatment during situations such as the use of contrast agents;
11. History of adverse events leading to permanent discontinuation of immunotherapy; or a history of grade 2 or higher immune-related pneumonitis or myocarditis;
12. Active or suspected autoimmune disease. Patients with autoimmune-related hypothyroidism who are undergoing thyroid hormone replacement therapy are permitted to participate in the study; patients with controlled Type 1 diabetes mellitus receiving insulin therapy are also allowed to participate in the study;
13. Live vaccinations or attenuated live vaccinations should not be administered within 4 weeks prior to the initial dosing. Administration of inactivated viral vaccines for seasonal influenza is permitted;
14. Known history of severe allergic reactions to macromolecular protein preparations/monoclonal antibodies, or allergy to components of the trial drug formulation；previous treatment with antibody-drug conjugates (ADCs) using a topoisomerase I inhibitor as the payload;
15. Active tuberculosis;
16. Human immunodeficiency virus (HIV) infection;
17. Pregnant or lactating women;
18. The researcher deems that the subject has any other factors that make them unsuitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-01-26 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-06-05 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 24 week
  Objective response rate (ORR) (assessed by INV according to the RECIST v1.1 criteria)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 14 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by INV according to the RECIST v1.1 criteria.

SECONDARY OUTCOMES:
ORR | up to 24 weeks
  Objective response rate (ORR) (assessed by the IRRC according to the RECIST v1.1 criteria)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 14 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by the IRRC according to the RECIST v1.1 criteria.
OS | From randomization to death from any cause (up to approximately 36 months)
  Overall Survival
Incidence and severity of adverse events (AEs) | time from the date of the first dose of study drug until the date of death from any cause, assessed up to 24 months
  severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version [v] 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, Dr., Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital, Jinan, Shandong, China